CLINICAL TRIAL: NCT03306615
Title: Peripheral Modulation of Muscle Stiffness and Spasticity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sheikh Khalifa Stroke Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00273264
Record Dates: First submitted 2017-10-03; First posted 2017-10-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Muscle Spasticity
Keywords: Muscle Stiffness; Muscle Spasticity; Stroke; Cerebral Palsy; Hyperreflexia
MeSH Terms: conditions — Muscle Spasticity; Stroke; Cerebral Palsy; Reflex, Abnormal | interventions — Hyaluronoglucosaminidase; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Hyaluronidase plus saline
  Interventions: Drug: Hyaluronidase
- Control Arm (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hyaluronidase — HYLENEX recombinant, diluted with 0.9% Sodium Chloride Injection
  Other Names: Hylenex
  Arms: Treatment Arm
Drug: Placebo — 0.9% Sodium Chloride Injection
  Other Names: Normal saline
  Arms: Control Arm

SUMMARY:
This is a single-center, double-blind, randomized, placebo-controlled, sequential Phase II trial of human recombinant hyaluronidase injections in individuals with post-stroke upper limb muscle stiffness. The investigators will recruit 56 subjects, who will be randomized to receive either the intervention or normal saline injections (first injection), and then the intervention the participants did not receive first (second injection). All individuals will receive the treatment by the end of the study.

DETAILED DESCRIPTION:
1. To test the effect of hyaluronidase injections on upper limb outcomes. The investigators will test the hypothesis that compared to placebo, human recombinant hyaluronidase injections will increase passive range of motion (ROM) in the most affected joint of the upper limb (primary outcome), isometric muscle strength or force generation capacity using Maximum Voluntary Contraction (MVC) on electromyography (EMG), reduce upper limb motor impairment as measured by the Fugl-Meyer (FM) scale, and improve function as measured by the Wolf Motor Function Test (WMFT).
2. To evaluate the effect of hyaluronidase on neural and non-neural components of muscle stiffness. The investigators will test the hypothesis that compared to placebo, intramuscular (IM) hyaluronidase will modulate the passive and potentially also the active component of the stretch reflex, reduce stiffness and improve arm motor control.
3. To determine the effect of hyaluronidase on intramuscular glycosaminoglycans (GAG) content. The investigators will test the hypothesis that compared to placebo, IM hyaluronidase will reduce the T1rho relaxation times in the biceps and triceps muscles of the affected arm.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke 4-180 months prior
* Moderately-severe muscle stiffness
* Lack of full passive and active range of motion in at least 2/4 areas (shoulder, elbow, forearm, wrist) in the hemiparetic upper limb;
* Willingness to have MRI, complete all clinical assessments, and comply with study protocols;
* Ability to give informed consent and HIPPA certifications; and

Exclusion Criteria:

* treatment of spasticity with Botulinum toxin or intrathecal baclofen within the past six months, phenol injections within the past 12 months, or ongoing adjustment of anti-spastic medications;
* other neurologic condition that may affect motor response (e.g., Parkinson's disease, amyotrophic lateral sclerosis (ALS), MS);
* clinically significant cognitive dysfunction with score <19 on Folstein's Mini Mental Status Examination or depression with score >10 on the Patient Health Questionnaire-9 (PHQ-9);
* pregnancy;
* known hypersensitivity to hyaluronidase;
* claustrophobia;
* standard contraindications for MRI
* Any condition that will preclude the patient from completing the protocol as determined by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Most affected upper limb joint passive range of motion (Cohort 1) | 9 weeks
  passive range of motion in most affected joint across the upper limb
Most affected upper limb joint passive range of motion (Cohort 2) | 15 weeks
  passive range of motion in most affected joint across the upper limb

SECONDARY OUTCOMES:
Total upper limb passive and active range of motion | 15 weeks
  passive and active range of motion in shoulder, elbow and forearm joints
Change in upper limb Fugl-Meyer Assessment Score | 15 weeks
  measures motor impairment in the affected upper limb, Score range is 0-66, and a higher score indicates a better outcome
Change in Wolf-Motor Function Test (WMFT) Score | 15 weeks
  Measures upper extremity function following stroke, Includes 6 items, with a 0-5 score range for each item, and a higher score indicates a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ning Cao, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States